CLINICAL TRIAL: NCT06305052
Title: Effects of Olfactory and Gustatory Stimulus on the Nutrition of Premature Babies: Double-blind Randomized Clinical Trial
Brief Title: Effects of Olfactory and Gustatory Stimulus on the Nutrition of Premature Babies
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Fernando Figueira Integral Medicine Institute (Other)
Responsible Party: Principal Investigator, João Guilherme Bezerra Alves, Principal Investigator, Professor Fernando Figueira Integral Medicine Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: estimulation-taste-olfactory; 65635922.0.0000.5201 (Other: CAAE (Certificate of Presentation of Ethical Review))
Record Dates: First submitted 2024-02-09; First posted 2024-03-12 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Weight, Birth; Premature Birth
Keywords: Nutrition; Prematurity; human milk; smell and taste
MeSH Terms: conditions — Birth Weight; Premature Birth; Anosmia | interventions — Milk; Water

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Milk group (Experimental): Olfactory and gustatory stimuli with milk in premature infants before tube feeding.
  Interventions: Other: Milk
- Placebo group (Placebo Comparator): Olfactory and taste stimuli with double-distilled water in premature infants before tube feeding
  Interventions: Other: Water

INTERVENTIONS:
Other: Milk — Premature newborns allocated to the intervention group will receive olfactory and taste stimuli immediately before feeding through an oral/nasal gastric tube.
  In the intervention group, the taste stimulus will be carried out through a drop of milk administered directly to the tongue of the premature baby if he is awake, if the newborn is sleeping the milk will be placed on his lips.
  The olfactory stimulus will be offered through a drop of milk using a cotton swab, positioned close to the premature baby's nostrils as close as possible without touching them, immediately before the tube diet.
  Arms: Milk group
Other: Water — In the control group, the taste stimulus will be done through a drop of double-distilled water on a cotton swab, then administered directly to the tongue of the premature baby if he is awake, however, when he is sleeping, the drop of water will be deposited on his lips. The olfactory stimulus in the control group will be carried out with a drop of double-distilled water using a cotton swab, positioned close to the nostrils as close as possible without touching them, immediately before carrying out the tube diet.
  Arms: Placebo group

SUMMARY:
The objective of this clinical trial is to test the effects of olfactory and taste stimulation with milk or water in premature newborns with a gestational age between 28 and 32 weeks.

The main question researchers want to resolve is: • Does olfactory and gustatory stimulation in these newborns reduce the time spent with an oral or nasogastric feeding tube and bring forward oral feeding? Participants will be stimulated with milk or water depending on the randomly chosen group. 1: the olfactory stimulus (with smell) will be performed with a sterile cotton swab close to the nostrils immediately before feeding through the tube, 2: the gustatory stimulus (taste) will be performed with a sterile cotton swab on which a drop of milk or water will be applied on the newborn's tongue if they are awake or on their lips if they are sleeping, and is performed immediately before tube feeding.

DETAILED DESCRIPTION:
The objective of this clinical trial is to test the effects of olfactory and taste stimulation with milk or water in premature newborns with a gestational age between 28 and 32 weeks.

Prematurity is the main cause of infant morbidity and mortality in Brazil. Nutritional problems caused by digestive immaturity are generally associated with undesirable outcomes in preterm infants, both immediate and late, and improving preemies' tolerance to milk has been challenging. The cephalic phase of digestion plays a crucial role in nutrient absorption. However, although it is known that smell and taste develop during intrauterine life, olfactory and taste stimuli have not yet been properly studied in the nutrition of premature babies. Objectives: to determine the effects of olfactory and gustatory stimuli on the nutrition of premature infants admitted to the neonatal intensive care unit of the Instituto de Medicina Integral Prof. Fernando Figueira (IMIP).Methods: a double-blind randomized clinical trial will be carried out in premature infants receiving enteral feeding via an oro/nasogastric tube. The study will be carried out at the IMIP university hospital, Recife-Pernambuco. The population will be composed of premature babies with a gestational age between 28 and 32 weeks and/or weighing < or equal to 1,500g and who are indicated for feeding through a naso/orogastric tube. The intervention will consist of olfactory and taste stimuli through breast milk. The primary outcome will be considered the period defined in days from the beginning of stimulation until the removal of the nasal or orogastric tube. Secondary outcomes will be considered: weight gain and anthropometric parameters, such as weight, length and head circumference at discharge from the NICU, as well as feeding time via oral/nasal and parenteral gastric tube, type of feeding at the time of secretion (natural or artificial) and diagnosis of necrotizing enterocolitis. The study is characterized as a prospective randomized clinical trial, with a pragmatic sample size determined during the recruitment period established at 10 months. Analysis will be performed by intention to treat. This project must be previously approved by the IMIP Ethics Committee and all participants must have their parents sign the Free and Informed Consent Form

ELIGIBILITY:
Inclusion Criteria:

* Newborns with Gestational Age (GA) between 28 and 32 weeks and/or birth weight ≤1,500g.
* Use of oro/nasogastric tube.

Exclusion Criteria:

* Newborns who have already started enteral feeding
* Twin newborns
* Congenital malformation associated with the digestive system that requires surgery soon after birth.
* Congenital conditions that impair growth

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Comparison of the period between the beginning of the intervention and enteral feeding. | until the moment when the newborn's oral or nasal gastric tube will be removed (evaluated up to 1 month).
  Comparison of the period between the beginning of the intervention and the completion of enteral feeding (removal of the oral or nasogastric tube), verified through the number of days in the period. will be verified in the newborn's medical record.

SECONDARY OUTCOMES:
Describe the gestational age of the newborn | until the moment of data collection from the medical records, which is equivalent to 1 day.
  This information will be collected from the newborn's medical record. Data regarding the gestational age of the newborn will be expressed in weeks.
Describe the sex of the newborn. | until the moment of data collection from the medical records, which is equivalent to 1 day.
  This information will be collected from the newborn's medical record. Data regarding the sex of the newborn will be expressed as female or male.
Describe the type of birth. | until the moment of data collection from the medical records, which is equivalent to 1 day.
  This information will be collected from the newborn's medical record. Data regarding the type of birth will be expressed as vaginal or cesarean section.
Describe the APGAR score. | until the moment of data collection from the medical records, which is equivalent to 1 day.
  This information will be collected from the newborn's medical record. The data regarding the APGAR score will be expressed in positive natural numbers from 0 to 10 in the first and fifth minutes of the newborn's life.
Describe birth weight and birth weight z-score. | until the moment of data collection from the medical records, which is equivalent to 1 day.
  The data will initially be checked in the medical record to obtain anthropometric parameters at birth: weight will be expressed in grams. The data obtained will be used in the Fenton 2013 calculator tool to obtain the zscores.
Describe head circumference at birth and head circumference z-score at birth | until the moment of data collection from the medical records, which is equivalent to 1 day.
  The data will initially be checked in the medical record to obtain anthropometric parameters at birth: the head circumference will be expressed in centimeters. The data will then be used in the Fenton 2013 calculator tool to obtain zscores.
Describe birth length and birth length z-score. | until the moment of data collection from the medical records, which is equivalent to 1 day.
  The data will initially be checked in the medical record to obtain anthropometric parameters at birth: length will be expressed in centimeters. The data will then be used in the Fenton 2013 calculator tool to obtain the zscores.
Determine the frequency of rupture of membranes >24h, chorioamnionitis, antepartum hemorrhage, gestational hypertension, pre-eclampsia and prenatal steroids >24h. | at the time of data collection from the medical record, which is equivalent to 1 day.
  This information will be collected from the newborn's medical record. They will be noted on a specific form created by the researchers to demonstrate, through alternatives between yes or no, the presence of these variables.
Compare the time, in days, of feeding via oral/nasal gastric tube. | until the moment the tube feeding time will be recorded in days (evaluated up to 2 months).
  The number of days that the newborn was fed through a tube will be recorded, using data provided in the medical record.
Compare the total duration, in days, of parenteral nutrition (TPN) use. | until the moment the time of parenteral nutrition feeding will be recorded in days (evaluated up to 15 days).
  The number of days that the newborn was fed by parenteral nutrition will be recorded, using data provided in the medical record.
Compare the type of food at discharge (natural, artificial or mixed). | until the moment when the type of food offered to the newborn upon discharge will be recorded (evaluated within 2 months).
  The type of food that the newborn received during hospital discharge will be presented, whether it was natural with breast milk, artificial with the use of milk formulas or mixed when premature, it received both types of food. They will be obtained through data in the medical record.
Compare weight gain and weight Z score, at 28 days of life and at discharge from the neonatal ICU, as well as anthropometric parameters: head circumference and length with their respective Z score at discharge from the NICU. | until the newborn is 28 days old (assessed until the 28th) and at discharge (up to 2 months)
  The data will initially be checked in the medical record to obtain anthropometric parameters: weight in grams, length in centimeters and head circumference in centimeters. The data will then be used in the Fenton 2013 calculator tool to obtain zscores.
Compare gestational age (GA) at the time of removal of the oro/nasogastric tube and at discharge from the NICU. | until removal of the newborn's tube (assessed up to 2 months) and at discharge (up to 2 months)
  The gestational age data referring to the moment the newborn's tube was removed and at the time of discharge will be expressed in weeks. This data will be collected from the medical record.
Compare the frequency of diagnosis of patent ductus arteriosus requiring treatment, bronchopulmonary dysplasia (BPD), retinopathy of prematurity, intraventricular hemorrhage and necrotizing enterocolitis. | until the moment of discharge of the newborn (evaluated up to 2 months).
  This information will be collected from the newborn's medical record. They will be noted on a specific form prepared by the researchers to demonstrate, through alternatives between yes or no, the presence of these variables.
Determine the association of treatment time with oxygen therapy (nasal catheter, nasal prong - nasal CPAP, intermittent positive pressure or endotracheal ventilation) in hours. | until the moment of discharge of the newborn (assessed up to 2 months).
  The medical record will check the treatment time in days, the treatment with oxygen therapy, whether it be (nasal catheter, nasal prong - nasal CPAP, intermittent positive pressure or endotracheal ventilation). After obtaining this data, the time will be transformed into hours and recorded on a specific research form.

CONTACTS AND LOCATIONS:
Overall Officials: João GB Alves, PhD, Study Director — Instituto de Medicina Integral Fernando Figueira IMIP; Luana GR Fonseca, Principal Investigator — Instituto de Medicina Integral Fernando Figueira IMIP
Locations (1):
- Instituto de Medicina Integral Professor Fernando Figueira, Recife, Pernambuco, Brazil